CLINICAL TRIAL: NCT00036582
Title: Clozapine vs Placebo In Treatment-Refractory Bipolar Disorder In Children And Adolescents
Brief Title: Clozapine vs. Placebo in Treatment-Refractory Bipolar Disorder in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020198; 02-M-0198
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-02

CONDITIONS: Bipolar Disorder
Keywords: Psychophysiology; Structural MRI; Genetics; Bipolar Disorder; Children and Adolescents; Clozapine; Placebo; Treatment-Refractory; Bipolar; Healthy Volunteer; HV; BPD; Normal Control
MeSH Terms: conditions — Bipolar Disorder | interventions — Clozapine

INTERVENTIONS:
Drug: Clozapine

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of clozapine in children and adolescents with treatment resistant bipolar disorder. This study will also explore how the brain functions in early-onset bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder (BPD) in children and adolescents is a serious illness that carries a high risk for chronicity, impairing comorbidities, and completed suicide. Treatment options are often limited by inefficacy or intolerable side effects. Open trials in adult bipolar subjects and several case series in children and adolescents provide preliminary evidence that clozapine, an atypical antipsychotic, may be effective in treatment-resistant bipolar disorder. The first specific aim of this study is to test the efficacy and safety of clozapine compared to placebo in a double-blind study of children and adolescents with treatment refractory BPD. Other specific aims involve exploring the pathophysiology of early-onset BPD by 1) testing the hypotheses that, compared to controls, children with BPD have increased psychophysiological reactivity to emotional stimuli and decreased prepulse inhibition; 2) obtaining samples of genetic material from affected probands and their parents for later analysis; and 3) identifying anatomic changes in the brains of children with BPD using structural MRI.

ELIGIBILITY:
INCLUSION CRITERIA (All 5 must be met): Children with BPD

Ages 8-17

Currently meets criteria for bipolar disorder, manic or mixed, as determined by the K-SADS diagnostic interview.

Treatment-resistant, defined as a history of unsuccessful trials of lithium (documented level of greater than 0.8 mEq/L), valproic acid (documented level of greater than 50 ug/ml), carbamazepine (documented level greater than or equal to 6 ug/ml), a neuroleptic as well as a combination of two of these agents. Each trial must have been at least 6 weeks long. A trial will be considered unsuccessful if the medication was discontinued because of intolerable side-effects.

The child should be in treatment with a community psychiatrist to whom they will return upon completion of the study.

Current CGAS score less than 50

EXCLUSION CRITERIA: Children with BPD

Full scale IQ less than 80

Meets criteria for substance use disorder in the three months prior to randomization

Currently pregnant, lactating, or sexually active without using a barrier method of contraception

Previous treatment with clozapine

History of seizures

History of leukopenia or agranulocytosis

Presence of an unstable medical illness

INCLUSION CRITERIA: CONTROLS

Control subjects will be age- and sex- matched to the BPD subjects. They will have normal physical and neurological examinations, and an identified primary care physician. Both control subjects and their first-degree relatives must be free of current or past psychopathology.

EXCLUSION CRITERIA: CONTROLS

I.Q less than 80; ongoing medical illness; neurologic disorder (including seizures); pregnancy; meeting past or present criteria for any diagnosis on the K-SADS-PL; meeting criterion A of post-traumatic stress disorder (exposure to a traumatic event).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116
Dates: Start 2002-05; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wozniak J, Biederman J, Kiely K, Ablon JS, Faraone SV, Mundy E, Mennin D. Mania-like symptoms suggestive of childhood-onset bipolar disorder in clinically referred children. J Am Acad Child Adolesc Psychiatry. 1995 Jul;34(7):867-76. doi: 10.1097/00004583-199507000-00010. PMID 7649957
- [Background] Geller B, Sun K, Zimerman B, Luby J, Frazier J, Williams M. Complex and rapid-cycling in bipolar children and adolescents: a preliminary study. J Affect Disord. 1995 Aug 18;34(4):259-68. doi: 10.1016/0165-0327(95)00023-g. PMID 8550951
- [Background] Faedda GL, Baldessarini RJ, Suppes T, Tondo L, Becker I, Lipschitz DS. Pediatric-onset bipolar disorder: a neglected clinical and public health problem. Harv Rev Psychiatry. 1995 Nov-Dec;3(4):171-95. doi: 10.3109/10673229509017185. PMID 9384947